CLINICAL TRIAL: NCT02959437
Title: A Phase 1/2 Study Exploring the Safety, Tolerability, Effect on the Tumor Microenvironment, and Efficacy of Azacitidine in Combination With Pembrolizumab and Epacadostat in Subjects With Advanced Solid Tumors and Previously Treated Stage IIIB or Stage IV Non-Small Cell Lung Cancer and Stage IV Microsatellite-Stable Colorectal Cancer (ECHO-206)
Brief Title: Azacitidine Combined With Pembrolizumab and Epacadostat in Subjects With Advanced Solid Tumors (ECHO-206)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-206 / ECHO-206; 2016-004289-25 (EudraCT Number)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors; Advanced Malignancies; Metastatic Cancer
Keywords: Solid tumors; NSCLC; CRC
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Azacitidine; pembrolizumab; epacadostat; INCB057643; INCB059872

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A: Azacitidine + Pembrolizumab + Epacadostat (Experimental): Part 1 is an open-label 3 + 3 + 3 dose-escalation design based on observing each dose level for a period of 21 days. Part 2 will evaluate the recommended dose determined in Part 1.
  Interventions: Drug: Azacitidine; Drug: Pembrolizumab; Drug: Epacadostat
- Treatment Group B: INCB057643 + Pembrolizumab + Epacadostat (Experimental): Part 1 is an open-label 3 + 3 + 3 dose-escalation design based on observing each dose level for a period of 42 days. Part 1 will also contain dose-expansion cohorts in previously treated NSCLC and MSS CRC. Part 2 will evaluate the recommended dose determined in Part 1.
  Interventions: Drug: INCB057643; Drug: Pembrolizumab; Drug: Epacadostat
- Treatment Group C: INCB059872 + Pembrolizumab + Epacadostat (Experimental): Part 1 is an open-label 3 + 3 + 3 dose-escalation design based on observing each dose level for a period of 42 days. Part 1 will also contain dose-expansion cohorts in previously treated NSCLC and MSS CRC. Part 2 will evaluate the recommended dose determined in Part 1.
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat; Drug: INCB059872

INTERVENTIONS:
Drug: Azacitidine — Five doses of azacitidine will be administered by subcutaneous injection or intravenously (IV) over Days 1 to 7 in Cycles 1 through 6.
  Arms: Treatment Group A: Azacitidine + Pembrolizumab + Epacadostat
Drug: Pembrolizumab — Pembrolizumab will be administered in a 30-minute IV infusion every 3 weeks on Day 1 of each 21-day cycle.
  Arms: Treatment Group A: Azacitidine + Pembrolizumab + Epacadostat
Drug: Epacadostat — Epacadostat tablets will be administered orally twice daily.
  Arms: Treatment Group A: Azacitidine + Pembrolizumab + Epacadostat
Drug: INCB057643 — INCB057643 will be orally self- administered once daily beginning on Cycle 1 Day 1 and continuously thereafter in 21-day cycles.
  Arms: Treatment Group B: INCB057643 + Pembrolizumab + Epacadostat
Drug: Pembrolizumab — Pembrolizumab will be administered in a 30-minute IV infusion every 3 weeks of each 21-day cycle starting on Cycle 2 Day 1.
  Arms: Treatment Group B: INCB057643 + Pembrolizumab + Epacadostat; Treatment Group C: INCB059872 + Pembrolizumab + Epacadostat
Drug: Epacadostat — Epacadostat tablets will be administered orally twice daily starting at Cycle 2 Day 1.
  Arms: Treatment Group B: INCB057643 + Pembrolizumab + Epacadostat; Treatment Group C: INCB059872 + Pembrolizumab + Epacadostat
Drug: INCB059872 — INCB059872 will be orally self- administered once daily OR every other day beginning on Cycle 1 Day 1 and continuously thereafter in 21-day cycles.
  Arms: Treatment Group C: INCB059872 + Pembrolizumab + Epacadostat

SUMMARY:
This is an open-label, Phase 1/2 study in subjects with advanced or metastatic solid tumors. The study has three separate treatment groups where separate epigenetic agents are evaluated with an immunotherapy combination. Treatment Group A will evaluate the DNA methyltransferase inhibitor azacitidine in combination with the programmed death receptor-1 (PD-1) inhibitor pembrolizumab and the indoleamine 2,3-dioxygenase (IDO-1) inhibitor epacadostat; Treatment Group B will evaluate the bromodomain and extra-terminal (BET) inhibitor INCB057643 with pembrolizumab and epacadostat; and Treatment Group C will evaluate the lysine-specific demethylase 1A (LSD1) inhibitor INCB059872 with pembrolizumab and epacadostat. The study will be divided into 2 parts (Part 1 and 2). Part 1 is a dose-escalation assessment to evaluate the safety and tolerability of the combination therapies. Once the recommended doses have been determined, subjects with previously treated NSCLC, microsatellite-stable colorectal cancer (CRC), head and neck squamous cell carcinoma, urothelial carcinoma, and melanoma will be enrolled into expansion cohorts in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written informed consent for the study.
* Willingness to undergo a pretreatment and on-treatment tumor biopsy to obtain tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Part 1: Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors that have failed prior standard therapy (disease progression; subject refusal or intolerance is also allowable).
* Part 2:

  *Note: Subjects must have failed available therapies that are known to confer clinical benefit as indicated below, unless they are ineligible, intolerant, or refused standard treatment.
* Subjects with histologically or cytologically confirmed NSCLC:

  * Metastatic (Stage IV) or recurrent NSCLC (according to American Joint Committee on Cancer 7th edition guidelines) who have had disease progression after available therapies for advanced or metastatic disease that are known to confer clinical benefit, been intolerant to treatment, or refused standard treatment.
  * Prior systemic regimens must include previously approved therapies, including a platinum-containing chemotherapy regimen; a tyrosine kinase inhibitor for tumors with driver mutations; and checkpoint inhibitors where approved.
  * Must have disease progression on a prior PD-1-pathway targeted agent.
* Subjects with recurrent (unresectable) or metastatic CRC:

  * Have histologically confirmed microsatellite stable (MSS) CRC.
  * Stage IV MSS CRC (according to American Joint Committee on Cancer 7th edition guidelines) who have had disease progression after available therapies for advanced or metastatic disease that are known to confer clinical benefit, been intolerant to treatment, or refused standard treatment.
  * Prior systemic regimens must include previously approved therapies, including fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy; an anti-VEGF therapy (if no contraindication); and if negative for KRAS, NRAS, and BRAF mutations and no contraindication, an anti-epidermal growth factor receptor (EGFR) therapy; and progressed after the last administration of approved therapy.
* Subjects with HNSCC:

  * Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
  * Carcinomas of the nasopharynx, salivary gland, or nonsquamous cell histology are excluded.
  * Must have received prior treatment with a platinum-based therapy
  * Must have had documented disease progression while on a prior PD-1 pathway-targeted agent.
* Subjects with melanoma:

  * Histologically or cytologically confirmed melanoma.
  * Unresectable Stage III or Stage IV melanoma, as per American Joint Committee on Cancer staging system not amenable to local therapy.
* Subjects with urothelial carcinoma:

  * Histologically or cytologically confirmed urothelial carcinoma of the renal pelvis, ureter, urinary bladder, or urethra that is transitional cell or mixed transitional/nontransitional (predominantly transitional) cell type.
  * Stage IV locally advanced or metastatic urothelial carcinoma (according to American Joint Committee on Cancer 7th edition guidelines) with documented disease progression while on a PD-1 pathway targeted therapy.

Exclusion Criteria:

* Laboratory parameters not within the protocol-defined range.
* Receipt of anticancer medications or investigational drugs within a defined interval before the first administration of study drug.
* Has not recovered from toxic effects of prior therapy to ≤ Grade 1.
* Active or inactive autoimmune disease or syndrome.
* Active infection requiring systemic therapy.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful.
* Has received a live vaccine within 30 days of planned start of study therapy.
* Prior receipt of an IDO inhibitor.
* Subjects with uncontrolled type I or type II diabetes mellitus (defined as HgbA1c > 8).
* Prior receipt of a BET inhibitor (Treatment Group B only).
* Subjects with a history of bleeding related to cancer under study requiring a medical intervention (eg, embolization procedure, RBC transfusion, or hospitalization) within 30 days of study enrollment (Treatment Groups B and C only).
* Clinically significant bleeding within 14 days of Cycle 1 Day 1 (Treatment Groups B and C only).
* Prior receipt of an LSD1 inhibitor including INCB059872 (Treatment Group C only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Hayer, MD, Study Director — Incyte Corporation
Locations (12):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego, La Jolla, California
  - The University of Chicago, Chicago, Illinois
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Sarah Cannon, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Spain (2):
  - Vall D Hebron Univ, Barcelona
  - Univ De Navarra, Pamplona
- United Kingdom (2):
  - University College London Hospitals (Uclh), London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 study sites in United States, 2 sites in UK and 1 site in Spain.
Pre-assignment Details: A total of 70 participants were enrolled in the study. Study enrollment was permanently discontinued on 15-Feb-2019 as a strategic decision. No patients were enrolled in Treatment Group B and Treatment Group C.
Groups:
- Treatment Group A :100mg of INCB24360: In Treatment Group A, subjects will receive the DNMT inhibitor azacitidine in combination with the PD-1 inhibitor pembrolizumab and the IDO1 inhibitor epacadostat at 100mg. Due to early termination of study subjects from dose escalation and dose expansion are combined.
- Treatment Group A :300mg of INCB24360: In Treatment Group A, subjects will receive the DNMT inhibitor azacitidine in combination with the PD-1 inhibitor pembrolizumab and the IDO1 inhibitor epacadostat at 300mg.
- Treatment Group B :INCB057643+Pembrolizumab+Epacadostat: In Treatment Group B, subjects will receive INCB057643 in combination with the PD-1 inhibitor pembrolizumab and the IDO1 inhibitor epacadostat at 100mg.
- Treatment Group C :INCB059872+Pembrolizumab+Epacadostat: In Treatment Group C, subjects will receive INCB059872 in combination with the PD-1 inhibitor pembrolizumab and the IDO1 inhibitor epacadostat at 100mg.
Period: Overall Study
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Started | 62 | 8 | 0 (Due to early termination of the trial Treatment groups B and C were not dosed.) | 0 (Due to early termination of the trial Treatment groups B and C were not dosed.)
Completed | 0 | 0 | 0 | 0
Not Completed | 62 | 8 | 0 | 0
Not completed — Death | 33 | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 3 | 0 | 0
Not completed — Progressive Disease | 9 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 0 | 0 | 0
Not completed — Other Unspecified | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled in Treatment Group B and C.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat | Total
Number analyzed (Participants) | 62 | 8 | 0 | 0 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.92) | 53.0 (11.31) |  |  | 56.5 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 4 |  |  | 23
  Male | 43 | 4 |  |  | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 56 | 5 |  |  | 61
  Black/African-American | 3 | 0 |  |  | 3
  Asian | 2 | 0 |  |  | 2
  American-Indian/Alaska Native | 0 | 0 |  |  | 0
  Native Hawaiian/Pacific Islander | 0 | 0 |  |  | 0
  Other | 1 | 3 |  |  | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino: Hispanic or Latino | 4 | 2 | 0 | 0 | 6
  Hispanic or Latino: Not Hispanic or Latino | 54 | 6 | 0 | 0 | 60
  Hispanic or Latino: Unknown | 4 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and 2 : Number of Participants With Treatment Emergent Adverse Events
Description: A treatment-emergent AE was defined as an event occurring after exposure to at least 1 dose of study drug. A treatment-related AE was defined as an event with a definite, probable, or possible causality to study medication. A serious AE is an event resulting in death, hospitalization, persistent or significant disability/incapacity, or is life threatening, a congenital anomaly/birth defect or requires medical or surgical intervention to prevent 1 of the outcomes above. The intensity of an AE was graded according to the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 4.03: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (life-threatening).
Time Frame: Baseline through 42-49 days after end of treatment, estimated up to 27 months (24 months with 100 day FU period).
Population: The safety population includes all subjects enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Number analyzed (Participants) | 62 | 8 | 0 | 0
Participants | 62 | 8 |  |

2. Primary Outcome: Part 1 and 2: Objective Response Rate Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. A participant was considered as an objective responder if the participant had a best overall response of CR or PR.
Time Frame: Every 9 weeks for the duration of study participation; estimated minimum of 6 months.
Population: The response evaluable population includes all subjects enrolled in the study who received at least 1 dose of study drug, completed a baseline scan and have at least 1 post baseline scan, or has been on study for a minimum of 70 days of follow-up or who discontinued treatment. No participants enrolled in part 2 of the study due to early termination of study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Number analyzed (Participants) | 62 | 8 | 0 | 0
Participants | 3 | 1 | 0 | 0

3. Secondary Outcome: Parts 1 and 2: Percentage of Responders Determined by Immunohistochemistry
Description: Responder is defined as an increase in the number of tumor-infiltrating lymphocytes or the ratio of CD8+ lymphocytes to T regulatory cells infiltrating tumor post-treatment versus pretreatment with pembrolizumab and epacadostat in combination with azacitidine.
Time Frame: Baseline to Week 5/6 or week 8/9
Population: All subjects enrolled in the study who received at least 1 dose of study drug, who had evaluable baseline and on treatment biopsies. No participants enrolled in part 2 of the study due to early termination of study.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group A :100 or 300mg of INCB24360: Treatment Group A :100mg of INCB24360 In Treatment Group A, subjects will receive the DNMT inhibitor azacitidine in combination with the PD-1 inhibitor pembrolizumab and the IDO1 inhibitor epacadostat at 100mg or 300mg. Due to early termination of study subjects from dose escalation and dose expansion are combined.
Arm/Group | Treatment Group A :100 or 300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Number analyzed (Participants) | 19 | 0 | 0
Participants
  Intratumoral CD8+ T cells | 14 |  |
  CD8+:FoxP3+ ratios | 10 |  |

4. Secondary Outcome: Parts 1 and 2: Progression-free Survival Based on RECIST v1.1.
Description: Defined as the time from date of first dose of study drug until the earliest date of disease progression per RECIST v1.1, or death due to any cause, if occurring sooner than progression.
Time Frame: Every 9 weeks from date of randomization until the date of first documented progression or date of death from any cause whichever came first, assessed up to 24 months
Population: All subjects enrolled in the study who received at least 1 dose of study drug, completed a baseline scan and have at least 1 post baseline scan, or has been on study for a minimum of 70 days of follow-up or who discontinued treatment. No participants enrolled in part 2 of the study due to early termination of study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Number analyzed (Participants) | 62 | 8 | 0 | 0
Months | 2.07 [1.97 to 2.17] | 2.64 [1.31 to 6.11] |  |

5. Secondary Outcome: Parts 1 and 2: Duration of Response Based on RECIST v1.1
Description: Defined as the time from earliest date of disease response until the earliest date of disease progression per RECIST v1.1, or death due to any cause, if occurring sooner than progression.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360 | Treatment Group B :INCB057643+Pembrolizumab+Epacadostat | Treatment Group C :INCB059872+Pembrolizumab+Epacadostat
Number analyzed (Participants) | 3 | 1 | 0 | 0
Months | 2.63 [2.20 to 21.85] | 1.22 [NA to NA] — Upper and Lower bound not estimable due to 1 responder in the treatment arm. |  |

ADVERSE EVENTS:
Time Frame: Baseline through 42-49 days after end of treatment, estimated up to 27 months (24 months with 100 day FU period).
Description: The safety population included all participants enrolled in the study who received at least 1 dose of study drug. Data is presented for Group A only, no participants enrolled in Treatment Groups B and C.
Arm/Group | Treatment Group A :100mg of INCB24360 | Treatment Group A :300mg of INCB24360
All-Cause Mortality (participants affected / at risk) | 41/62 | 4/8
Serious Adverse Events (participants affected / at risk) | 28/62 | 3/8
Other Adverse Events (participants affected / at risk) | 59/62 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A :100mg of INCB24360 (N=62) | Treatment Group A :300mg of INCB24360 (N=8)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinua tachycardia (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 1
Disease Progression (General disorders) | 8 | 0
Fatigue (General disorders) | 2 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Urinary tract Infection (Infections and infestations) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Wound Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Injury (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysmetria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Confusional State (Psychiatric disorders) | 1 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A :100mg of INCB24360 (N=62) | Treatment Group A :300mg of INCB24360 (N=8)
Anaemia (Blood and lymphatic system disorders) | 11 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 12 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 16 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 34 | 3
Vomiting (Gastrointestinal disorders) | 21 | 2
Chills (General disorders) | 4 | 1
Fatigue (General disorders) | 28 | 6
Injection site erythema (General disorders) | 5 | 0
Injection site pain (General disorders) | 4 | 0
Injection site reaction (General disorders) | 13 | 0
Local swelling (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 6 | 1
Pyrexia (General disorders) | 6 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 3
Blood alkaline phosphatase increased (Investigations) | 7 | 2
Blood creatinine increased (Investigations) | 4 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Headache (Nervous system disorders) | 4 | 4
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 5 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Pneumaturia (Renal and urinary disorders) | 0 | 1
Terminal dribbling (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Hypotension (Vascular disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT02959437/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02959437/SAP_000.pdf